CLINICAL TRIAL: NCT03934138
Title: Does the Subject's Understanding of Underlying Placebo Mechanisms Compensate for the Loss of Efficacy Associated With the Disclosure of the Use of a Placebo
Brief Title: Does the Understanding of Placebo Mechanisms Compensate for the Loss of Efficacy Associated With Open Label Placebo
Acronym: PLACETHIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoire TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A01643-50
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Acute Pain
Keywords: Placebo; Experimental pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: 2 groups : Educated open label placebo And Conventional placebo
  Each of the subjects will undergo the Cold Pressure text procedure under the condition of interest and a control.
Who Masked: Participant
Masking Description: Only the subjects in the the conventional placebo group will be masked. In the educated open label placebo group, subjects will be aware that the cream is inert.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educated open label placebo (Active Comparator): These subjects will undergo all the same procedures as in the control group. But before the placebo CTP, they will watch a short movie explaining placebo mechanisms. While applying the placebo cream, they will be told that the cream is inert (placebo), efficient to decrease pain caused by cold and the mechanisms seen in the movie will take place.
  Interventions: Other: Educational movie on placebo mechanisms
- Conventional placebo (Placebo Comparator): These subjects will watch a video on hand washing. While applying the placebo cream, they will be told that this cream is effective to decreased pain caused by cold.
  Interventions: Other: Informative movie on hand washing

INTERVENTIONS:
Other: Educational movie on placebo mechanisms — Educational movie on placebo mechanisms : animated video, duration : 12 minutes.
  It will be followed by the CPTs : experimentally induced pain by keeping the non dominant hand in cold water (1° Celsius) for a limited time. The duration of immersion is personal and calibrated to be around to ensure that the intensity of pain will be homogeneous (around 7/10 on the visual analogue scale with no treatment)
  Other Names: Cold Pressure Test (CPT)
  Arms: Educated open label placebo
Other: Informative movie on hand washing — Animated video, duration : 11 minutes. It will be followed by the CPTs : experimentally induced pain by keeping the non dominant hand in cold water (1° Celsius) for a limited time. The duration of immersion is personal and calibrated to be around to ensure that the intensity of pain will be homogeneous (around 7/10 on the visual analogue scale with no treatment).
  Other Names: Cold Pressure Test (CPT)
  Arms: Conventional placebo

SUMMARY:
The investigators are investigating whether, when given detailed information about underlying placebo mechanisms and pain, subjects will have a response similar to that of those subjected to a procedure in which they receive a conventional placebo treatment (associated with deception).

STUDY DESIGN: This is a non-inferior parallel, controlled and randomized, single blind trial.

POPULATION: The investigators will include in the study 126 subjects without known pathology. Participants will then be divided into 2 groups on a randomized basis.

METHODOLOGY: Each subject will undergo three sessions of Cold Pressure Test (CPT), a cold pain stimulation method: calibration, condition of interest (conventional placebo or educated placebo) and control. The investigators' main judgment criterion is be the difference in pain intensity experienced on the visual analog scale between the CPT control and the CPT under the condition of interest.

This study will allow the investigators to rule on the non-inferiority of an educated open label placebo compared to a conventional placebo in the context of an acute painful stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated to Social Security
* Informed consent, written and signed by the subject.

Exclusion Criteria:

* Persons referred to in Articles L1121-5 to L1121-8 of the Public Health Code (CSP), which corresponds to all protected persons: pregnant women, parturient women, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons subject to a legal protection measure, cannot be included in clinical trials.
* Persons with a pathology against indicating the use of CPT experimentally induced pain :
* Any pathologies affecting the venous, arterial or lymphatic system
* Diabetes
* Cardiac disorders
* Asthma
* Frostbite
* Epilepsy
* Arthritis
* Lupus erythematosus
* Allergy to Cremafluid® cream
* Person with concomitant treatment that modifies sensitivity to pain, chronic or acute at the time of the experiment, such as analgesics, psychotropic drugs or anti-inflammatories.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-05-03 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: Visual Analogue Scale (VAS) | At the end of the CPT procedure, within 30 seconds after the removal of the hand from the CPT cold water tank.
  Evaluated with a Visual Analogue Scale (VAS) from 0 to 100 mm, with a non inferiority margin at 10 mm and a standard deviation at 22 mm.

SECONDARY OUTCOMES:
Anxiety respiratory frequency change | During the CPT procedure
  Evaluated thanks to the respiratory frequency collect with a PneumoTrace belt through LabChart software.
Anxiety blood pressure change | During the CPT procedure
  Evaluated thanks to the automatic blood pressure monitor (both systolic/diastolic blood pressure, heart rate)
Knowledge of placebo's mechanisms | At the beginning and end of the CPT procedures
  Evaluated with a questionnaire made for this study with 17 questions about placebo mechanisms.
Perception of the investigator | At the end of the study, when all CPT procedures have been carried out, within 10 minutes after the last immersion
  The perception of the investigator will be evaluated by a visual analogue scale "perception of the investigator".
The Perceived Awareness of the Research Hypothesis Scale questionnaire | At the end of the study, when all CPT procedures have been carried out, within 10 minutes after the last immersion
  Perception of the research hypothesis with the Rubin Questionnaire. Perceived Awareness of the Research Hypothesis " (PARH) wich is a scale of 4-item quantitative self-report method for measuring the potential influence of demand characteristics in research situations

OTHER OUTCOMES:
Blood pressure | About 1 minute before every CPT procedures and within 10 secondes after each CPT procedures
  Safety measure to insure blood pressure does not exceed 150/90mmHg (both systolic/diastolic blood pressure, heart rate)

CONTACTS AND LOCATIONS:
Overall Officials: Leo DRUART, Principal Investigator — TIMC IMAG Thémas team; SaraEve GRAHAM LONGSWORTH, Principal Investigator — TIMC IMAG Thémas team; Nicolas PINSAULT, Study Director — TIMC IMAG Thémas team
Locations (2):
- France (2):
  - Leo Druart, Grenoble
  - Saraeve Graham Longsworth, Grenoble

REFERENCES:
- [Background] Kaptchuk TJ, Friedlander E, Kelley JM, Sanchez MN, Kokkotou E, Singer JP, Kowalczykowski M, Miller FG, Kirsch I, Lembo AJ. Placebos without deception: a randomized controlled trial in irritable bowel syndrome. PLoS One. 2010 Dec 22;5(12):e15591. doi: 10.1371/journal.pone.0015591. PMID 21203519
- [Background] Locher C, Frey Nascimento A, Kirsch I, Kossowsky J, Meyer A, Gaab J. Is the rationale more important than deception? A randomized controlled trial of open-label placebo analgesia. Pain. 2017 Dec;158(12):2320-2328. doi: 10.1097/j.pain.0000000000001012. PMID 28708766
- [Background] Benedetti F, Carlino E, Pollo A. How placebos change the patient's brain. Neuropsychopharmacology. 2011 Jan;36(1):339-54. doi: 10.1038/npp.2010.81. Epub 2010 Jun 30. PMID 20592717
- [Background] Benedetti F, Amanzio M. Mechanisms of the placebo response. Pulm Pharmacol Ther. 2013 Oct;26(5):520-3. doi: 10.1016/j.pupt.2013.01.006. Epub 2013 Jan 28. PMID 23370213
- [Background] Colloca L, Howick J. Placebos Without Deception: Outcomes, Mechanisms, and Ethics. Int Rev Neurobiol. 2018;138:219-240. doi: 10.1016/bs.irn.2018.01.005. Epub 2018 Apr 4. PMID 29681327
- [Background] Voudouris NJ, Peck CL, Coleman G. The role of conditioning and verbal expectancy in the placebo response. Pain. 1990 Oct;43(1):121-128. doi: 10.1016/0304-3959(90)90057-K. PMID 2277714
- [Background] Pecina M, Zubieta JK. Expectancy Modulation of Opioid Neurotransmission. Int Rev Neurobiol. 2018;138:17-37. doi: 10.1016/bs.irn.2018.02.003. Epub 2018 Apr 2. PMID 29681324
- [Background] Mitchell LA, MacDonald RA, Brodie EE. Temperature and the cold pressor test. J Pain. 2004 May;5(4):233-7. doi: 10.1016/j.jpain.2004.03.004. PMID 15162346
- [Background] Streff A, Kuehl LK, Michaux G, Anton F. Differential physiological effects during tonic painful hand immersion tests using hot and ice water. Eur J Pain. 2010 Mar;14(3):266-72. doi: 10.1016/j.ejpain.2009.05.011. Epub 2009 Jun 21. PMID 19540783
- [Background] Carvalho C, Caetano JM, Cunha L, Rebouta P, Kaptchuk TJ, Kirsch I. Open-label placebo treatment in chronic low back pain: a randomized controlled trial. Pain. 2016 Dec;157(12):2766-2772. doi: 10.1097/j.pain.0000000000000700. PMID 27755279
- [Derived] Druart L, Graham Longsworth S, Rolland C, Dolgopoloff M, Terrisse H, Bosson JL, Pinsault N. Can an Open-Label Placebo Be as Effective as a Deceptive Placebo? Methodological Considerations of a Study Protocol. Medicines (Basel). 2020 Jan 2;7(1):3. doi: 10.3390/medicines7010003. PMID 31906435